CLINICAL TRIAL: NCT06818955
Title: Clinical Study on the Safety and Efficacy of Orlistat in Third-generation EGFR-TKI Resistance
Brief Title: Orlistat Overcoming Third-generation EGFR-TKI Resistance
Acronym: OOTER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ping Peng (Other)
Collaborators: Hubei Cancer Hospital (Other)
Responsible Party: Sponsor-Investigator, Ping Peng, PhD，MD，Principal Investigator，Department of Thoracic Oncology, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGFR-TKI resistance study
Record Dates: First submitted 2025-02-03; First posted 2025-02-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Lung Adenocarcinoma; Osimertinib
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Orlistat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- orlistat group (Experimental): For patients who are resistant to osimertinib and require continued oral administration of targeted drugs, we will add orlistat
  Interventions: Drug: Orlistat 120 mg

INTERVENTIONS:
Drug: Orlistat 120 mg — Orlistat 120 mg po tid

SUMMARY:
EGFR mutation positivity accounts for 50% of lung adenocarcinoma cases. Multiple clinical trials, represented by FLAURA, AENEAS, and FURLONG studies, have confirmed that third-generation EGFR-TKI can provide significant benefits to patients with EGFR sensitive mutations and has become the first-line preferred treatment for EGFR mutation positive NSCLC, with a median PFS of around 19 and OS of around 38 months. These large-scale Phase III studies have confirmed the excellent efficacy of third-generation EGFR-TKI in EGFR mutation positive patients. However, regardless of the targeted drug, resistance will occur within less than 2 years. Blood test data for first-line treatment with osimertinib showed that the most common forms of resistance were secondary MET amplification (20%), EGFR C797S mutation (8%), PIK3CA, Her-2 amplification, and so on. The mechanism of resistance is complex and has many factors. Currently, for the treatment of third-generation EGFR-TKI resistance, the IMPOWER150 and ORIENTAL31 treatment modes are commonly used. Although the combination of these four drugs has good efficacy, the side effects are significant. Some patients are unwilling to undergo chemotherapy due to physical problems and hope to continue taking targeted drugs orally. Orlistat is a long-acting and potent specific gastrointestinal lipase inhibitor that can directly block the absorption of body fat. It is commonly used for weight loss in clinical practice and is relatively inexpensive. Our project team found in vitro and in vivo data that orlistat can effectively promote sensitivity to osimertinib. The combination of orlistat and osimertinib can overcome osimertinib resistance without significant toxic side effects. For patients who are unwilling to undergo chemotherapy and require continued oral targeted therapy, the investigators attempted to add orlistat to see if it can improve resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Previously received three generations of systemic TKI treatment and developed resistance (including Axitinib, Amitinib, Fumatinib, Bevatinib, Lazetinib, etc.);
2. General condition score ECOG 0-2 points;
3. Expected survival period of more than 3 months;
4. Laboratory examination:

   ① WBC≥3.5×109／L，ANC≥1.5×109／L，PLT≥80×109／L， Hb≥90g/L；

   ② Blood BUN and creatinine are within 1.5 times the upper limit of normal values;

   ③ TBIL ≤ 1.5 times the upper limit of normal value;

   ④ ALT and AST ≤ 2.5 times the upper limit of normal values; Patients with liver metastasis should not exceed 5 times the upper limit of normal values;

   ⑤ Normal coagulation function (PT, APTT within 1.5 times the upper limit of normal range).
5. The patient requests to continue taking targeted drugs orally
6. Voluntarily sign the informed consent form, with expected compliance.

Exclusion Criteria:

1. Suffering from serious medical diseases, including serious heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, serious infection, and active gastrointestinal ulcer;
2. A large amount of pleural and pericardial effusion requires immediate treatment;
3. Brain metastases with clinical symptoms;
4. Pregnant or lactating women;
5. The patient is able to tolerate chemotherapy and is willing to accept it

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-16 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of cycle 3 (each cycle is 21 days)
  Overall response rate (ORR) was defined as the combination of CR and PR.

SECONDARY OUTCOMES:
Safety (Rate of grade 3 and higher grade treatment-related adverse events) | From date of treatment allocation until treatment completion 30 days
  Adverse events will be evaluated and recorded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0)

IPD SHARING:
Plan to Share IPD: No